CLINICAL TRIAL: NCT04423146
Title: Advanced Methods for Improving Anesthesiologic Management and Their Effect on Perioperative Outcome in Scoliosis Surgery, Especially in Childhood (SCOL Study): a Prospective Observational Study
Brief Title: Anesthesiologic Management Effect on Perioperative Outcome in Scoliosis Surgery
Acronym: SCOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, assoc.prof.MD,Ph.D, Brno University Hospital
Other Study IDs: SCOL 2020
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Scoliosis
Keywords: scoliosis; surgery; scoliosis surgery; Motor evoked potentials
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients scheduled for elective scoliosis surgery: Patients scheduled for elective scoliosis surgery will be anesthetized in TIVA mode,combining propofol and remifentanil with titration to the target BIS value. Motor evoked potentials will be measured and evaluated by members of operating team perioperatively. The quality of evoked potentials (poor vs good quality) and the actual value of amplitude and latency at different BIS levels (40 - 60) will be monitored.
  Interventions: Other: The evocation of reproducible motor evoked potential according to the different BIS levels

INTERVENTIONS:
Other: The evocation of reproducible motor evoked potential according to the different BIS levels — The evocation of reproducible motor evoked potential and the actual value of amplitude and latency at different BIS levels (40 - 60) will be monitored.

SUMMARY:
Alteration of evoked potentials is described in cases with using inhalation anaesthetics. Muscle relaxants are contraindicated in case of motor evoked potentials except for initial dose for intubation of the patient. Dominant anaesthetic method for procedures with measuring motor evoked potentials is total intravenous anaesthesia (TIVA). Bispectral index (BIS) monitoring is one of the possible options for comprehensive monitoring of the depth of general anaesthesia. It helps to optimize the management of anaesthesia, so it reduces the risk of perioperative awakenings due to shallow anaesthesia or inadequate depth of anaesthesia associated with the risk of cognitive dysfunction, as well as investigators expect worse interpretation of motor evoked potentials. At the same time, it shortens the time to wake up from general anaesthesia after hours-long surgery. BIS monitoring allows optimizing the depth of anaesthesia and leads to improve quality and interpretation of motor evoked potentials. The depth of TIVA managed by BIS affects the reproducibility of motor evoked potentials.

DETAILED DESCRIPTION:
SCOL study is designed as a prospective observational study. We will monitor patients with scoliosis suitable for TIVA with BIS monitoring after the approval by the ethical committee of the University Hospital Brno and the Faculty of Medicine of Masaryk University in Brno, Czech Republic. The study period is planned from 1st September 2020 to 31st December 2024. Anaesthesia will be maintained following standardized local protocol for scoliosis surgery, include preoperative preparation and premedication. General anaesthesia will be performed in TIVA mode,combining propofol and remifentanil with titration to the target BIS value. Motor evoked potentials will be measured and evaluated by members of operating team perioperatively. The evocation of reproducible motor evoked potential and the actual value of amplitude and latency at different BIS levels (40 - 60) will be monitored. Motor evoked potentials (MEP) reproducibility will be based on standardized orthopaedic practice, according to the amplitude, latency of the MEP. The reproducibility will be monitored in defined surgery phases: before skin incision at the different BIS levels, next after screw application, rod applications, after distraction and the last one before wound suturing. At the same time, the BIS value is recorded.

In addition to the MEP reproducibility, investigators will measure the amplitude and latency value. These parameters and actual BIS value will be monitored in each patient after the recovery from neuromuscular blockade (TOF ratio value above 90%) to eliminate the influence of neuromuscular blockade on neurophysiology monitoring. Due to individual variability in the MEP latency and amplitude in these patients, the initial MEP value will be set as the default (100%), and other values will be expressed as a percentage.

Other monitored parameters in this study will be blood loss, blood derivates and transfusion products administered to the patient in first 24 hours after surgery, the time between the end of the surgery and extubation, neurological complications, number of surgical revisions and a total length of hospitalization.

The annual number of scoliosis operations at the University hospital Brno is around 130 patients. It is the largest surgery centre in Central Europe.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for scoliosis surgery with perioperative MEP monitoring

Exclusion Criteria:

* Scoliosis surgery without perioperative MEP monitoring
* Contraindication for perioperative MEP monitoring
* Contraindication of using propofol (soy, egg lecithin or peanuts allergy,...) or other drugs used for anaesthesia
* The inability of attachment of BIS electrodes to the standard position

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients indicated for elective scoliosis surgery with perioperative MEP monitoring
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The evocation of reproducible motor evoked potentials at different BIS levels (40 - 60) | During the scoliosis surgery
  The evocation of reproducible motor evoked potentials at different BIS levels (40 - 60) will be monitored according to standardized orthopaedic practise for evaluation of MEP.

SECONDARY OUTCOMES:
MEP parameters | During the scoliosis surgery
  MEP parameters (latency and amplitude) parameters will be monitored in defined surgery phases with recording the actual MEP values and BIS value after recovery from neuromuscular blockade. The initial MEP value will be set as the default (100%), and other values will be expressed as a percentage. We will analyze scoliosis subgroups, the idiopathic and neuromuscular scoliosis.

OTHER OUTCOMES:
Perioperative blood management | 24 hours postoperatively
  blood loss, blood derivates and transfusion products administered to the patient in first 24 hours after surgery
Surgical complications | 30 days postoperatively
  Neurological complications and number of surgical revisions within 30 days and length of days of hospitalization will be recorded.
Anaesthesiology management data | Intraoperative period until extubation
  Surgery length, the interval between the end of surgery to extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Repko Martin, prof. MD., Ph.D., Study Chair — Faculty of medicince Masaryk University and University Hospital Brno
Locations (1):
- Faculty hospital Brno, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided